CLINICAL TRIAL: NCT00742235
Title: hCAP18 Levels and Vitamin D Deficiency in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ishir Bhan, MD, MPH, Instructor in Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-0003000/1
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Subjects; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vitamin D insufficient (treated with ergocalciferol 50,000 IU every other day x 5 doses)
  Interventions: Drug: ergocalciferol
- Vitamin D sufficient (No Intervention): Subjects who did not receive ergocalciferol and had a 25-OH vitamin D level >32 ng/ml

INTERVENTIONS:
Drug: ergocalciferol — Ergocalciferol 50,000 IU given every other day for 5 total doses
  Other Names: Vitamin D
  Arms: 1

SUMMARY:
Vitamin D deficiency (low levels of vitamin D in the blood) is a common problem. A recently discovered protein, called hCAP18, likely plays an important role in the immune system and may depend on adequate levels of vitamin D. It is not known what levels of vitamin D are needed to allow the body to make this protein. Nor is it known if giving vitamin D to people who are found to be deficient will help boost levels of hCAP18. This study aims to clarify the relationship between vitamin D levels and hCAP18.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80

Exclusion Criteria:

* Known active infectious disease or chronic inflammatory disorder
* Hypercalcemia
* Chronic kidney disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ishir Bhan, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited via flyer to a clinical research center.
Pre-assignment Details: Subjects were excluded for eGFR<60, hypercalcemia, history of nephrolithiasis.
Groups:
- Vitamin D Sufficient: Subjects not treated with ergocalciferol and who had 25-OH vitamin D > 32 ng/ml.
- Vitamin D Insufficient: Subjects found to have an initial 25-OH vitamin D level < 32 ng/mL who were offered ergocalciferol 50,000 IU every other day x 5 doses (250,000 IU total)
Period: Overall Study
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient
Started | 32 | 67
Completed | 32 | 36
Not Completed | 0 | 31
Not completed — Lost to Follow-up | 0 | 31

BASELINE CHARACTERISTICS:
Groups:
- Vitamin D Sufficient: Subjects with baseline 25-OH vitamin D levels ≥ 32 ng/ml were not treated with ergocalciferol.
- Vitamin D Insufficient: Subjects found to have an initial 25-OH vitamin D level < 32 ng/mL were treated with ergocalciferol 50,000 IU every other day x 5 doses (250,000 IU total) and returned for repeat laboratory studies.
- Total: Total of all reporting groups
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient | Total
Number analyzed (Participants) | 32 | 67 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 66 | 98
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (14.9) | 36.7 (12.5) | 36.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 11 | 37 | 48
Region of Enrollment [Number; unit: participants]
  United States | 32 | 67 | 99

OUTCOME MEASURES:

1. Primary Outcome: hCAP18 Levels
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient
Number analyzed (Participants) | 29 | 65
ng/ml | 762 (347) | 639 (286)

2. Primary Outcome: Baseline 25-OH Vitamin D Level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient
Number analyzed (Participants) | 32 | 67
ng/ml | 40 [40 to 51.5] | 25 [20 to 29]

ADVERSE EVENTS:
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/36
Other Adverse Events (participants affected / at risk) | 0/0 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No